CLINICAL TRIAL: NCT05030350
Title: A Phase 3 Open-label Safety Trial of PH94B Nasal Spray in the Acute Treatment of Anxiety in Adult Subjects With Social Anxiety Disorder (SAD)
Brief Title: Open-label Safety Trial of PH94B in Social Anxiety Disorder (SAD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped by the sponsor for business reasons and not due to any safety concerns with PH94B
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH94B-CL030
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PH94B 3.2 micrograms (Experimental): 100 microliter nasal spray to each nostril up to four times a day as needed for acute anxiety
  Interventions: Drug: PH94B

INTERVENTIONS:
Drug: PH94B — Nasal spray

SUMMARY:
This study evaluates the safety and tolerability of PH94B with repeated dosing over a period of up to 12 months. Participating subjects will use PH94B up to 4 times a day when they encounter anxiety-provoking situations in daily life. Safety and tolerability of PH94B (≤ 4 doses per day up to 12 months) will be assessed and summarized during monthly visits from baseline (Visit 2) to end of treatment (Visit 14) in AEs, laboratory values, 12-lead ECGs, physical examinations, and vital sign assessments following exposure to PH94B.

ELIGIBILITY:
Most but not all patients will enter the study following completion of Palisade-1 (NCT047548020) and Palisade-2 (NCT05011396).

Inclusion Criteria:

1. Male and female adults, 18 through 65 years of age, inclusive.
2. Women of childbearing potential must be able to commit to the consistent and correct use of an effective method of birth control throughout the study, and must also have a negative urine pregnancy test result at both Screening (Visit 1) (for subjects who attend Visit 1) and Baseline (Visit 2), prior to IP administration. Effective methods of contraception include: condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), or implantable contraceptive devices.
3. Current diagnosis of social anxiety disorder
4. Clinician-rated HAM-D17 total score < 18 at study entry
5. LSAS score 50 or greater

Exclusion Criteria:

1. Any history of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, psychosis, anorexia or bulimia, autism-spectrum disorder, or obsessive-compulsive disorder. Any other current Axis I disorder, other than SAD, which is the primary focus of treatment. Note that subjects with concurrent Generalized Anxiety Disorder are eligible for the study provided that Generalized Anxiety Disorder is not the primary diagnosis.
2. Subjects who meet criteria for moderate or severe alcohol or substance use disorder within the 1 year prior to study entry.
3. In the opinion of the Investigator, the subject has a significant risk for suicidal behavior during the course of their participation in the study.
4. Clinically significant nasal pathology or history of significant nasal trauma, nasal surgery, total anosmia, or nasal septum perforation that may have damaged the nasal chemosensory epithelium.
5. An acute or chronic condition, including an infectious illness, uncontrolled seasonal allergies at the time of the study, or significant nasal congestion that potentially could affect drug delivery to the nasal chemosensory epithelium.
6. Subjects using the following psychotropic medications: anticonvulsants, mood stabilizers, antipsychotic medications, gabapentin, pregabalin, opioids, naltrexone, esketamine, and ketamine at enrollment.

   Subjects using lower doses of atypical antipsychotics at Screening may be eligible after discussion with the Medical Monitor (e.g., quetiapine < 100 mg).

   In general, subjects using antidepressants or buspirone can continue to receive these provided that they have been taking them for a minimum of 2 months, and have been on a stable dose for a minimum of 1 month.
7. Use of anxiolytics, such as benzodiazepines or unapproved treatments such as beta blockers, within 30 days before study entry; concomitant use is prohibited during the study. Subjects who have been taking benzodiazepines daily for 1 month or longer at the time of Visit 1 are not eligible to participate.
8. Use of any over-the-counter product, prescription product, or herbal preparation for treatment of the symptoms of anxiety or social anxiety within 30 days before study entry; concomitant use is prohibited during the study.
9. Subjects with clinically significant abnormalities in hematology, blood chemistry, urinalysis, 12-lead ECG, or physical examination identified at the Screening visit or Baseline visit that in the clinical judgment of the Investigator, could place the subject at undue risk, interfere with study participation, or confound the results of the study.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaakko Lappalainen, MD, PhD, Study Director — VistaGen Therapeutics
Locations (3):
- United States (3):
  - VistaGen Investigational Site, Watertown, Massachusetts
  - VistaGen Investigational Site, New York, New York
  - VistaGen Investigational Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PH94B 3.2 Micrograms: PH94B Nasal Spray - administration of 3.2 micrograms PH94B, as needed, up to four times per day.
Period: Overall Study
Arm/Group | PH94B 3.2 Micrograms
Started | 481
Completed | 0
Not Completed | 481
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 8
Not completed — Lost to Follow-up | 35
Not completed — Pregnancy | 2
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 60
Not completed — Study terminated by sponsor | 349
Not completed — Positive Drug Screen | 4
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Groups:
- PH94B: PH94B Nasal Spray - administration of 3.2 micrograms PH94B, as needed, up to four times per day.
Arm/Group | PH94B
Number analyzed (Participants) | 481
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 481
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300
  Male | 181
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 41
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 87
  White | 318
  More than one race | 13
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 481

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Subjects with at least one Serious Adverse Event (SAE)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PH94B
Number analyzed (Participants) | 481
Participants
  Subjects with at least one TEAE | 273
  Subjects with at least 1 Mild TEAE | 186
  Subjects with at least 1 Moderate TEAE | 78
  Subjects with at least 1 Severe TEAE | 9
  Subjects with at least 1 TEAE leading to study discontinuation | 14
  Subjects with at least 1 SAE | 6

2. Other Pre Specified Outcome: Change in Total Liebowitz Social Anxiety Scale (LSAS) Scores Over Time With Use of PH94B
Description: The LSAS is a clinician-rated scale that has been shown to be sensitive to treatment-related change in social anxiety symptoms. The scale consists of 24 items. Each item is given 2 ratings: fear or anxiety on scale of 0 to 3 (with 0 = none and 3 = severe) and avoidance on a scale of 0 to 3 (with 0 = never and 3 = usually), with a total maximum overall score of 144. The sum of the 24 fear or anxiety items and the sum of the 24 avoidance items are combined for a total LSAS score.
Time Frame: V 2 (Baseline), V 3 (Month 1), V 4 (Month 2), V 5 (Month3), V 6 (Month 4), V 7 (Month 5), V 8 (Month 6), V 9 (Month 7), V 10 (Month 8), V11 (Month 9)
Population: The number analyzed differs from overall number analyze as PH94B-CL030 was terminated early by the sponsor
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PH94B
Number analyzed (Participants) | 480
score on a scale
  Visit 2 (Baseline) | 93.4 (18.79)
  Visit 3 (Month 1): number analyzed (Participants) | 385
  Visit 3 (Month 1) | 76.6 (24.63)
  Visit 4 (Month 2): number analyzed (Participants) | 324
  Visit 4 (Month 2) | 73.0 (25.09)
  Visit 5 (Month 3): number analyzed (Participants) | 218
  Visit 5 (Month 3) | 67.6 (25.58)
  Visit 6 (Month 4): number analyzed (Participants) | 164
  Visit 6 (Month 4) | 66.0 (24.85)
  Visit 7 (Month 5): number analyzed (Participants) | 119
  Visit 7 (Month 5) | 64.8 (24.91)
  Visit 8 (Month 6): number analyzed (Participants) | 85
  Visit 8 (Month 6) | 65.2 (23.70)
  Visit 9 (Month 7): number analyzed (Participants) | 53
  Visit 9 (Month 7) | 61.1 (26.44)
  Visit 10 (Month 8): number analyzed (Participants) | 26
  Visit 10 (Month 8) | 54.0 (21.52)
  Visit 11 (Month 9): number analyzed (Participants) | 7
  Visit 11 (Month 9) | 54.4 (7.76)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | PH94B
All-Cause Mortality (participants affected / at risk) | 1/481
Serious Adverse Events (participants affected / at risk) | 6/481
Other Adverse Events (participants affected / at risk) | 137/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PH94B (N=481)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Suicide attempt (Psychiatric disorders) | 1
Pelvic abscess (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Diverticulitis intestinal perforated (Infections and infestations) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PH94B (N=481)
Headache (Nervous system disorders) | 82
COVID-19 (Infections and infestations) | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT05030350/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT05030350/SAP_001.pdf